CLINICAL TRIAL: NCT04029987
Title: Bilateral Ultrasound-Guided Intra Muscular Quadratus Lumborum Block Versus Trans Muscular Quadratus Lumborum Block for Peri-Operative Analgesia in Abdominal Surgeries in Pediatric Patients. A Comparative Controlled Randomized Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Eslam Ragab ElSayed Mohamed Heggy, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-31-2018
Record Dates: First submitted 2018-12-02; First posted 2019-07-23 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: age:5-12, American Society of Anesthesia I-III, abdominal laparoscopies, randomly allocated into one of the study groups, randomization sequence will be concealed in sealed envelopes with alphabetic codes. The identifiers will be attached to the opened envelopes and secured by dedicated person independent of randomization proceedings. Patients, parents and data analysts will be blinded to group assignments.
  The groups:
  * group A → Trans muscular quadrous lamborum block (n=22)
  * group B → Intra muscular quadrous lamborum block (n=22)
  * group c → control (n=22) will receive conventional analgesia. Sample size Starting number of 22 patients for each group, Recalculation of the sample size will be carried out after studying 10 patients per group.
  The alpha error is set at 0.05 and the study power is 0.95.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients, parents and data analysts will be blinded to group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trans Muscular Quadratus Lumborum fascial plane Block (Active Comparator): In group (Trans Muscular Quadratus Lumborum Block),will undergo ultrasound guided trans-muscular quadratus lamborum block as follows:
  A 22 G echogenic needle will be inserted in plane from the posterior (medial) end of the probe and directed for the fascial plane between the Quadratus Lumborum and the Psoas Major muscles through the Quadratus Lumborum muscle. Once the needle is confirmed in correct location, 1 mL of saline will be injected after negative aspiration. Then 0.5 mL/Kg per side of bupivacaine 0.25% will be injected. The spread of the injectate should be observed to distribute within this plane. This technique will be repeated to the other side.
  Interventions: Procedure: Bilateral Ultrasound-Guided Transmuscular Quadratus Lumborum Block.
- Intra Muscular Quadratus Lumborum fascial plane Block (Active Comparator): In group Intra Muscular Quadratus Lumborum Block ,will undergo ultrasound guided intra-muscular quadratus lamborum (QL) block as follows:
  A 22 G echogenic needle will be inserted in plane from ventral (lateral) edge of the probe and advanced until penetration of QL muscle fascia is observed. Once the needle is confirmed in correct location, 1 mL of saline will be injected after negative aspiration. Then 0.5 mL/Kg per side of bupivacaine 0.25% will be injected. The spread of the injectate should be observed to distribute within this plane. This technique will be repeated to the other side.
  Interventions: Procedure: Bilateral Ultrasound-Guided intra smuscular Quadratus Lumborum Block.
- group c → control (Placebo Comparator): group c → control ,will receive conventional analgesia in the form of paracetamol with 15 mg\ k.g every 6 hours, and naluphin 0.1 mg \kg on demands
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Bilateral Ultrasound-Guided Transmuscular Quadratus Lumborum Block. — A 22 G echogenic needle will be inserted in plane from the posterior (medial) end of the probe and directed for the fascial plane between the Quadratus Lumborum and the Psoa Major muscles through the Quadratus Lumborum muscle. Once the needle is confirmed in correct location, 1 mL of saline will be injected after negative aspiration. Then 0.5 mL/Kg of bupivacaine 0.25% will be injected. The spread of the injectate should be observed to distribute within this plane. This technique will be repeated to the other side.
  Arms: Trans Muscular Quadratus Lumborum fascial plane Block
Procedure: Bilateral Ultrasound-Guided intra smuscular Quadratus Lumborum Block. — A 22 G echogenic needle will be inserted in plane from ventral (lateral) edge of the probe and advanced until penetration of QL muscle fascia is observed. Once the needle is confirmed in correct location, 1 mL of saline will be injected after negative aspiration. Then 0.5 mL/Kg of bupivacaine 0.25% will be injected. The spread of the injectate should be observed to distribute within this plane. This technique will be repeated to the other side.
  Arms: Intra Muscular Quadratus Lumborum fascial plane Block
Procedure: Control — Conventional analgesia
  Arms: group c → control

SUMMARY:
To compare between the intra muscular quadratous lamborum and the Trans muscular quadratous lamborum in pediatric population under going abdominal surgeries regards to first request of rescue analgesia, degree of pain relief, effect on hemo dynamic stability and incidence of complications.

DETAILED DESCRIPTION:
The investigators hypothesized that an ultrasound guided quadratous lamborum block would prove successful peri-operative analgesia for abdominal surgeries in pediatric patients, and that Intra muscular quadratous lamborum is non inferior to Trans muscular blockade with the advantage of being safer (away from the peritoneum and retroperitoneal organs) and with the assumption that sarcolemmal layer in pediatrics should not resist the diffusion of the injectant from within the muscle out, to reach the inter fascial plane where the targeted nerves are found and cause an efficient blockade.

ELIGIBILITY:
Inclusion Criteria:

* Children age starting from 5 to 12 years.
* Genders eligible for study: both sexes.
* American Society Of Anesthesia (ASA) I-III.
* Scheduled to undergo laparoscopy.

Exclusion Criteria:

* Refusal of regional block or patients requiring emergency procedures.

  * Known Local Anesthetics drug sensitivity
  * Bleeding disorders with International Normalised Ratio (INR) > 1.5 and/or platelets < 100 000.
  * Skin lesions or wounds at site of proposed needle insertion.
  * Evidence of peritonitis or septicemia.
  * Hepatic disease or enlargement.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Time of the first postoperative analgesic request | starting 15 minutes post extubation, then at time intervals of 30 minutes , 60 minutes, 6 hours and 12 hours
  (duration of the block, time spent post-operative before rescue opioid is needed at pain score of 6 or higher, up to 12 hours post operative.

SECONDARY OUTCOMES:
total opioid consumption over the first 12 hours. | through out the first 12 hours post operative.
  rescue analgesia in the form of intravenous nalbuphine 0.1 milligram/Kilogram will be given for a Wong-Baker Faces Scale more than 4 up to 12 hours post operative.
Pain score up to 12 hours after surgery. | through out the first 12 hours post operative.
  Postoperative pain score for each patient will be assessed by Wong-Baker Faces Scale at the following intervals: 15, 30, and 60 min, 6, and 12 hours after surgery.
Block failure | through out the first hour post operative.
  a failed block is where the patient requires more than two doses of rescue analgesia in the first hour postoperatively
Ease of performance of each technique | through out the block performance time
  Easiness of performance of the technique, rated on a simple verbal scale easy/moderately difficult/difficult) and defined as follows:
  * Easy block: successful block after the 1st skin puncture.
  * Moderately difficult block: successful block after more than one puncture or with the need for needle redirection or image optimization (as adjustment of depth, gain, or focus to visualize the needle path)
  * Difficult block: successful block after more than one puncture and with the with the need for needle redirection and image optimization
Block performance time | starting from probe contact with skin till 30 minutes.
  Block performance time in minutes which is the time from probe contact with skin till needle withdrawal
The incidence of post block adverse effects | starting after the block is given up to the first 12 hours post operative
  incidence of complications, such as:
  * postoperative nausea and vomiting, urinary retention, lower limb weakness
  * injury to the underlying structures (injury to the liver or a viscus), or hematoma formation as recorded under ultrasound guidance
  * need of postoperative mechanical ventilation or ICU admission
  * LA toxicity.

OTHER OUTCOMES:
patient's heart rate | starting from 5 minutes after intubation till 30 minutes after extubation
  heart rate will be recorded at the following intervals: T0 (baseline); 5 minutes after intubation, T1; 1 minute after skin incision, T2; 15 minutes after skin incision, T3; 30 minutes after skin incision, T4; 60 minutes after skin incision, T5; 90 minutes after skin incision, T6; 5 minutes after extubation, T7; 30 minutes after extubation in the recovrery area.
patient's systolic blood pressure | starting from 5 minutes after intubation till 30 minutes after extubation
  systolic blood pressure will be recorded at the following intervals: T0 (baseline); 5 minutes after intubation, T1; 1 minute after skin incision, T2; 15 minutes after skin incision, T3; 30 minutes after skin incision, T4; 60 minutes after skin incision, T5; 90 minutes after skin incision, T6; 5 minutes after extubation, T7; 30 minutes after extubation in the recovrery area.
patient's diastolic blood pressure | starting from 5 minutes after intubation till 30 minutes after extubation
  diastolic blood pressure will be recorded at the following intervals: T0 (baseline); 5 minutes after intubation, T1; 1 minute after skin incision, T2; 15 minutes after skin incision, T3; 30 minutes after skin incision, T4; 60 minutes after skin incision, T5; 90 minutes after skin incision, T6; 5 minutes after extubation, T7; 30 minutes after extubation in the recovrery area.
intraoperative administration of extra analgesic dose of fentanyl | starting from 10 minutes after the chosen block is given till extubation.
  Number of patients in each group who needed intraoperative administration of extra analgesic dose of fentanyl 0.5 microgram/kilogram),in patients showing increase in heart rate and/or arterial blood pressure 10 minutes after returning to supine position after the block is given, by more than 20% of baseline values (5 minutes after intubation) in response to surgical stimulus or thereafter throughout the whole operation.
Duration of surgery | starting from skin incision up to skin closure.
  time in minutes from skin incision till skin closure
Duration of general anesthesia | starting from induction of anesthesia till extubation
  time in minutes from induction of GA till extubation

CONTACTS AND LOCATIONS:
Locations (1):
- Abu ElReesh hospital, Cairo university Hospital,Kasr Alini, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No